CLINICAL TRIAL: NCT02654782
Title: Lactated Ringer's Versus 5% Human Albumin: A Double-Blinded, Randomized, Prospective Study in Cardiac Surgical Patients
Brief Title: Lactated Ringer's Versus 5% Human Albumin: Cardiac Surgical Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Student performing study left Mayo Clinic, no funds to continue study.
Sponsor: William C. Oliver (Other)
Responsible Party: Sponsor-Investigator, William C. Oliver, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-000858
Record Dates: First submitted 2016-01-08; First posted 2016-01-13 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Hemodynamic Stability
Keywords: Lactated Ringer's; Human Albumin
MeSH Terms: interventions — Ringer's Lactate; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lactated Ringer's (Active Comparator): Subjects randomized to Lactated Ringer's for hemodynamic resuscitation. Volume will be decided based off of individual patient needs.
  Interventions: Drug: Lactated Ringer's
- 5% Human Albumin (Active Comparator): Subjects randomized to 5% human albumin for hemodynamic resuscitation. Volume will be decided based off of individual patient needs.
  Interventions: Drug: 5% Human Albumin

INTERVENTIONS:
Drug: Lactated Ringer's — Crystalloid fluid given for hemodynamic resuscitation based off of individual patient needs.
  Arms: Lactated Ringer's
Drug: 5% Human Albumin — Colloid given for hemodynamic resuscitation based off of individual patient needs.
  Arms: 5% Human Albumin

SUMMARY:
The purpose of this study is to show which of two different types of fluid is best for cardiac surgical patients. During and after the subject's heart surgery, the subject will be given either Lactated Ringer's or 5% human albumin to replace lost blood and body fluids and to regulate blood pressure.

Albumin (human) 5% is a sterile, liquid preparation of albumin derived from large pools of human plasma. All units of human plasma used in the manufacture of Albumin (human) 5% are provided by FDA approved blood establishments only.

Lactated Ringer's is a sterile, nonpyrogenic solution containing isotonic concentrations of electrolytes in water for injection. It is FDA approved for administration by intravenous infusion for parental replacement of extracellular losses of fluid and electrolytes.

The hypothesis of this study is that the individual total fluid volume and alveolar-arterial gradient will be less with 5% human albumin compared to Lactated Ringer's in the perioperative cardiac surgical patient.

DETAILED DESCRIPTION:
Following Institutional Review Board (IRB) approval and written informed patient consent, 40 elective, cardiac surgical patients will be randomized to two different fluid therapy regimens, 5% human albumin only or Lactated Ringer's only, beginning in the intraoperative period and up to 6 hours in the intensive care unit. Providers and patients will be blinded to the fluid administered in the operating room and intensive care unit. The primary outcome measure will be the total volume of 5% human albumin or Lactated Ringer's given during the study period to maintain specified hemodynamic guidelines. Hemodynamic instability will be defined according to each patient's stipulated baseline parameters. Fluid will be administered at the request of providers in the operating room and intensive care unit in compliance with a perioperative fluid algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant female patients
* Patients undergoing elective cardiac surgery
* Aspirin, heparin, or warfarin preoperatively accepted

Exclusion Criteria:

* Previous sternotomy
* Emergency surgery
* Combined procedures (vascular or thoracic operations)
* Congenital heart repair
* Hypothermic cardiopulmonary bypass (CPB) < 28 degrees C
* Serum creatinine greater than or equal to 1.5 mg/dL
* Dialysis dependent renal failure
* Neurologic injury or event within 30 days (including transient ischemic attack)
* Cerebrovascular accident with significant residual neurologic deficit
* Severe chronic obstructive pulmonary disease with Forced Expiratory Volume in 1 Second (FEV1) < 45% of predicted value
* Home oxygen use
* Previous difficult intubation
* Acute normovolemic blood conservation techniques
* Liver disease with serum aspartate aminotransferase (AST) > 31 U/L
* Circulatory arrest
* Thrombolysis
* Pre-existing clotting disorder
* Platelet receptor glycoprotein IIb/IIIa (GP IIb/IIIa) antagonist medication received within 48 hours
* Steroids
* Ejection Fraction < 40%
* Intra-aortic balloon pumps
* Ongoing congestive heart failure
* Ventricular assist devices
* Total hearts
* Pregnant women
* Adults lacking capacity to consent
* Any patients initially enrolled in the study that end up with an intra-aortic balloon pump, left ventricular assist device, or on extracorporeal membrane oxygenation will be eliminated from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Oliver, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Lactated Ringer's | 5% Human Albumin
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactated Ringer's | 5% Human Albumin | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 5 | 9
  Asian, Indian | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Fluid Administered Indexed to Weight
Description: Adequate fluid volume plays a major part in maintaining the necessary hemodynamics to prevent organ damage during cardiac surgery. This will be measured by the total volume of fluid administered to the subject from the start of surgery up to 6 hours in the intensive care unit.
Time Frame: Start of surgery up to 6 hours into the intensive care unit (ICU)
Population: The study was terminated early. This was a student project and the student performing the study left Mayo Clinic and there were no funds to continue study. Targeted enrollment of 40 subjects was not met and data was not analyzed.
Arm/Group | Lactated Ringer's | 5% Human Albumin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Alveolar-arterial Gradient
Description: Alveolar-arterial gradient will be calculated from arterial blood gases on each patient. This value will be used to compare shunt in each arm.
Time Frame: Calculated throughout the study up to 6 hours in the ICU
Population: as for outcome 1
Arm/Group | Lactated Ringer's | 5% Human Albumin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Approximately 6 hours after surgery.
Arm/Group | Lactated Ringer's | 5% Human Albumin
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The study was terminated early. This was a student project and the student performing the study left Mayo Clinic and there were no funds to continue study. Targeted enrollment of 40 subjects was not met and data was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02654782/Prot_SAP_000.pdf